CLINICAL TRIAL: NCT02065141
Title: Validation Of A New Method To Simultaneously Measure Protein Digestion And Absorption
Brief Title: Method To Measure Protein Digestion & Absorption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University (Other)
Responsible Party: Principal Investigator, Marielle PKJ Engelen, PhD, PhD, Texas A&M University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2013-0758F
Record Dates: First submitted 2013-11-26; First posted 2014-02-17 (Estimated); Last update posted 2022-02-07 (Actual); Status verified 2022-02

CONDITIONS: Chronic Heart Failure; Pulmonary Disorder, Chronic Obstructive
Keywords: digestion; absorption; protein; amino acids; heart failure; COPD
MeSH Terms: conditions — Lung Diseases; Heart Failure; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Healthy (Other): screening visit: body weight and composition by DXA, height, and vital signs will be assessed.
  study day: stable isotope infusions with blood draws, sip feed
  Interventions: Other: sip feeding with stable isotope infusion
- Chronic Obstructive Pulmonary Disorder (Other): screening visit: body weight and composition by DXA, height, and vital signs will be assessed. Subjects may sign a medical release form to obtain medical information about them that will help determine study eligibility or can be used for later coding.
  study day: stable isotope infusions with blood draws, sip feed
  Interventions: Other: sip feeding with stable isotope infusion
- Chronic Heart Failure (Other): screening visit: body weight and composition by DXA, height, and vital signs will be assessed. Subjects may sign a medical release form to obtain medical information about them that will help determine study eligibility or can be used for later coding.
  study day: stable isotope infusions with blood draws, sip feed
  Interventions: Other: sip feeding with stable isotope infusion

INTERVENTIONS:
Other: sip feeding with stable isotope infusion — such as glycerol, D2O, tyrosine, phenylalanine, glucose, arginine, and citrulline

SUMMARY:
The aim of the present study is to validate a new method in healthy volunteers and those diagnosed with COPD and CHF that is able to measure protein digestion and absorption simultaneously. This method is used to quantify digestion and absorption in patients who are suspect of impaired digestion and absorption resulting in loss of nutrients.Findings may be used to develop treatment strategies to improve protein digestion and absorption in these patient groups.

DETAILED DESCRIPTION:
The study involves 1 screening visit of approximately 1-2 hours and 1 test day of approximately 8 hours. On the study day protein digestion and absorption will be measured using a mixture of amino acids that are made slightly heavier than normal, called stable isotopes. Subjects will receive feeding by sips to monitor changes in digestion and absorption, which can be picked up by stable isotope technology.

ELIGIBILITY:
IInclusion and exclusion criteria for study participation:

We will enroll subjects (males and females of all races) based on the inclusion/exclusion criteria described below. All subjects should be able to walk, sit and stand up indepedently. Screening procedures will be done prior to the study.

Inclusion criteria - CHF subjects:

* Ability to walk, sit down and stand up independently
* Age 45 years or older
* Ability to lie in supine or elevated position for 9 hours
* Diagnosis of CHF; under regular care by cardiologist
* Reduced ejection fraction (<45%) assessed in the past 2 years
* NYHA class II-IV
* Clinically stable condition; no hospitalization 4 weeks preceding first study day
* Willingness and ability to comply with the protocol

Inclusion criteria - COPD subjects:

* Ability to walk, sit down and stand up independently
* Age 45 years or older
* Ability to lie in supine or elevated position for 8 hours
* Diagnosis of moderate to very severe chronic airflow limitation and compliant to the following criteria: FEV1 < 70% of reference FEV1
* Clinically stable condition and not suffering from a respiratory tract infection or exacerbation of their disease (defined as a combination of increased cough, sputum purulence, shortness of breath, systemic symptoms such as fever, and a decrease in FEV1 > 10% compared with values when clinically stable in the preceding year) at least 4 weeks prior to the first test day
* Shortness of breath on exertion
* Willingness and ability to comply with the protocol

Inclusion criteria - healthy subjects:

* Healthy male & female according to the investigator's or appointed staff's judgment
* Age 45 years and older, or 20 - 30 for healthy young group

Exclusion Criteria - all subjects:

* Any condition that may interfere with the definition 'healthy subject' according to the investigator's judgment (healthy subjects only)
* Established diagnosis of malignancy
* History of untreated metabolic diseases including hepatic or renal disorder
* Presence of acute illness or metabolically unstable chronic illness
* Presence of fever within the last 3 days
* Body mass index >40 kg/m2 (healthy subjects only)
* Any other condition according to the PI or nurse that was found during the screening visit, that would interfere with the study or safety of the patient
* Use of protein or amino acid containing nutritional supplements within 5 days prior first study day
* Current Use of long-term oral corticosteroids (CHF only)
* Use of short course of oral corticosteroids within 4 weeks preceding first study day
* Failure to give informed consent or Investigator's uncertainty about the willingness or ability of the subject to comply with the protocol requirements
* (Possible) pregnancy
* Already enrolled in another clinical trial and that clinical trial interferes with participating in this study

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2014-11; Primary Completion 2019-01-19 (Actual); Study Completion 2019-01-19 (Actual)

PRIMARY OUTCOMES:
protein metabolism in gut | In postabsorptive and prandial state every 20 minutes up to 8 hours before each sip feeding on study day
  Digestion of the stable tracers of amino acid measured by plasma samples

SECONDARY OUTCOMES:
Body Composition | on screening or study day 1
  Body composition as measured by Dual-Energy X-ray Absorptiometry
Respiratory muscle strength | on study day 1
  determined by measurement of maximum breathing pressures
Skeletal muscle strength of hand | 30 minutes on screening or study day
  measurement of handrip strenth
Skeletal muscle strength of leg | 30 minutes on screening or study day
  measurement of muscle strength of leg using kin-com machine

CONTACTS AND LOCATIONS:
Overall Officials: Nicolaas E Deutz, PhD, Principal Investigator — Texas A&M University; Marielle P Engelen, PhD, Principal Investigator — Texas A&M University
Locations (1):
- Texas A&M University, College Station, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Engelen MPKJ, Kirschner SK, Coyle KS, Argyelan D, Neal G, Dasarathy S, Deutz NEP. Sex related differences in muscle health and metabolism in chronic obstructive pulmonary disease. Clin Nutr. 2023 Sep;42(9):1737-1746. doi: 10.1016/j.clnu.2023.06.031. Epub 2023 Jul 26. PMID 37542951